CLINICAL TRIAL: NCT01063803
Title: An Open-Label Extension Study To Assess The Long-term Safety And Tolerability Of ATN-103 In Subjects With Rheumatoid Arthritis
Brief Title: Study Evaluating Long-Term Safety Of ATN-103 In Subjects With Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ablynx, a Sanofi company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3242K1-2003; B2271005
Record Dates: First submitted 2010-02-02; First posted 2010-02-05 (Estimated); Last update posted 2016-04-11 (Estimated); Status verified 2013-01

CONDITIONS: Rheumatoid Arthritis
Keywords: Open-label; Long-term safety study of ATN-103 in RA
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1: ATN-103_30mg (Experimental)
  Interventions: Drug: ATN-103
- Arm 2: ATN-103_80 mg (Experimental)
  Interventions: Drug: ATN-103

INTERVENTIONS:
Drug: ATN-103 — A single subcutaneous injection of ATN-103 every 4 weeks (approx 13 SC injections during the study)
  Arms: Arm 1: ATN-103_30mg
Drug: ATN-103 — A single subcutaneous injection of ATN-103 every 4 weeks (approx 13 SC injections during the study)
  Arms: Arm 2: ATN-103_80 mg

SUMMARY:
This open-label extension study will allow subjects who have completed either the 3242K1-2000-WW or 3242K1-2001-JA study to receive up to an additional 48 weeks of ATN-103 treatment and will provide data on the long-term safety and tolerability of ATN-103 in subjects with rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have completed study 3242K1-2000-WW or 3242K1-2001-JA and have had no events that, in the opinion of the investigator, would preclude entry or participation in this study.

Exclusion Criteria:

* Pregnant or nursing women.
* Any major illness/condition or evidence of an unstable clinical condition (eg, renal, hepatic, cardiovascular, hematological, gastrointestinal, endocrine, pulmonary, immunologic [eg, Felty syndrome, human immunodeficiency virus (HIV) infection], infectious, neurological, or cerebral psychiatric disease, or evidence of demyelinating disease) that, in the investigator's judgment, will substantially increase the risk associated with the subject's developing an adverse event (AE) or serious adverse event (SAE) during the study, or preclude the evaluation of the subject's response.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2010-02; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Collection of safety data and assessments will include adverse events, treatment-emergent adverse events, injection site reactions, infections, vital signs and safety laboratory measurements. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — Ablynx NV
Locations (65):
- United States (25):
  - Investigational Site, Birmingham, Alabama
  - Investigational Site, Huntsville, Alabama
  - Investigational Site, Peoria, Arizona
  - Investigational Site, Riverside, California
  - Investigational Site, Upland, California
  - Investigational Site, Bridgeport, Connecticut
  - Investigational Site, Newark, Delaware
  - Investigational Site, Ocala, Florida
  - Investigational Site, Port Orange, Florida
  - Investigational Site, Vero Beach, Florida
  - Investigational Site, Coeur d'Alene, Idaho
  - Investigational Site, Frederick, Maryland
  - Investigational Site, Lansing, Michigan
  - Investigational Site, Freehold, New Jersey
  - Investigational Site, Charlotte, North Carolina
  - Investigational Site, Winston-Salem, North Carolina
  - Investigational Site, Columbus, Ohio
  - Investigational Site, Oklahoma City, Oklahoma
  - Investigational Site, Tulsa, Oklahoma
  - Investigational Site, Lake Oswego, Oregon
  - Investigational Site, Columbia, South Carolina
  - Investigational Site, Myrtle Beach, South Carolina
  - Investigational Site, Nashville, Tennessee
  - Investigational Site, Dallas, Texas
  - Investigational Site, San Antonio, Texas
- Canada (5):
  - Investigational Site, Winnipeg, Manitoba
  - Investigational Site, Kitchener, Ontario
  - Investigational Site, St. Catharines, Ontario
  - Investigational Site, Toronto, Ontario
  - Investigational Site, Québec, Quebec
- Hungary (2):
  - Investigational Site, Budapest
  - Investigational Site, Debrecen
- Japan (19):
  - Investigational Site, Nitona-cho, Chuoh-ku, Chiba-shi, Chiba
  - Investigational Site, Bunkyoucho, Matsuyama, Ehime
  - Investigational Site, Chuoh-ku, Fukuoka-shi, Fukuoka
  - Investigational Site, Kurume, Fukuoka
  - Investigational Site, Yoshio-machi Iizuka-shi, Fukuoka
  - Investigational Site, Tohrimachi, Takasaki, Gunma
  - Investigational Site, Katō, Hyōgo
  - Investigational Site, Kumamoto, Kumamoto
  - Investigational Site, Honmachi, Higashiyama, Kyoto
  - Investigational Site, Miyazaki, Miyazaki
  - Investigational Site, Nagano, Nagano
  - Investigational Site, Yamato, Sasebo, Nagasaki
  - Investigational Site, Higashi-tyo, Kawachi Nagano, Osaka
  - Investigational Site, Ureshino-machi, Ureshino-shi, Saga-ken
  - Investigational Site, Kawagoe, Saitama
  - Investigational Site, Midori-cho 2 Chome Tokorozawa-shi, Saitama
  - Investigational Site, Kawada-cho, Shinjyuku-ku, Tokyo
  - Investigational Site, Shinanomachi, Shinjuku, Tokyo
  - Investigational Site, Takaoka-shi, Toyama
- Russia (7):
  - Investigational Site, Kemerovo
  - Investigational Site, Moscow
  - Investigational Site, Novosibirsk
  - Investigational Site, Orenburg
  - Investigational Site, Ryazan
  - Investigational Site, Vladimir
  - Investigational Site, Yaroslavl
- Serbia (2):
  - Investigational Site, Belgrade, Serbia
  - Investigational Site, Niška Banja
- South Africa (4):
  - Investigational Site, Les Marais, Gauteng
  - Investigational Site, Berea, KwaZulu-Natal
  - Investigational Site, Panorama, Western Cape
  - Investigational Site, Pinelands, Western Cape
- Investigational Site, Chur, Switzerland